CLINICAL TRIAL: NCT01673854
Title: A Single Arm Open-Label Phase II Study of Vemurafenib Followed by Ipilimumab in Subjects With Previously Untreated V600 BRAF Mutated Advanced Melanoma
Brief Title: Phase II Safety Study of Vemurafenib Followed by Ipilimumab in Subjects With V600 BRAF Mutated Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA184-240; 2012-002054-24 (EudraCT Number)
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg (Experimental): Participants received vemurafenib, 960 mg, twice daily for 6 weeks (Vem1 Phase). After a washout period of 3-10 days, patients received ipilimumab, 10 mg/kg, every 3 weeks for a maximum of 4 doses. At Week 24, participants received ipilimumab, 10 mg/kg, every 12 weeks until disease progression or unacceptable toxicity. Patients who did not progress or have unacceptable toxicity in the Vem1 Phase were retreated with vemurafenib (Vem 2 Phase) at the last dose level identified at the end of the Vem1 Phase until disease progression or unacceptable toxicity.
  Interventions: Drug: Ipilimumab; Biological: Vemurafenib

INTERVENTIONS:
Drug: Ipilimumab
  Other Names: Yervoy®; BMS-734016
Biological: Vemurafenib
  Other Names: Zelboraf®

SUMMARY:
The purpose of this study is to assess the safety profile of vemurafenib, 960 mg, administered for 6 weeks, followed by ipilimumab monotherapy in patients with BRAF V600 mutated advanced/metastatic melanoma.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Key Inclusion Criteria:

* Men and women 18 years of age and older
* Histologic diagnosis of malignant melanoma tested positive for the BRAF V600 mutation
* Previously untreated unresectable Stage III or Stage IV melanoma
* Complete set of brain/neck, chest, abdomen/pelvis axial radiographs taken within 28 days of first dose of study drug
* Measurable melanoma by physical or radiographic examination
* Brain metastases stable after radiation for at least 1 month and off corticosteroid therapy for ≥30 days prior to enrollment
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Adequate hematologic parameters and renal and hepatic function

Key Exclusion Criteria:

* Primary ocular melanoma
* Active brain metastases with symptoms or requiring corticosteroid treatment
* Any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* History of or current active autoimmune diseases, including but not limited to inflammatory bowel diseases, rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis, systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies
* History of or current immunodeficiency disease, splenectomy, or splenic irradiation
* Prior anticancer therapy or investigational products <4 weeks prior to enrollment
* Prior therapy with a BRAF or MEK inhibitor and prior investigational anticancer immunotherapies;
* Prior therapies with immunosuppressive agents within the past 2 years
* Concomitant therapy with any anticancer or potent immunosuppressive agent, surgery, radiotherapy, other investigational anticancer therapies, or chronic use of systemic corticosteroids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-09-13 (Actual); Primary Completion 2014-07-25 (Actual); Study Completion 2015-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (14):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Baptist Cancer Institute, Jacksonville, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University Of New Mexico Cancer Center, Albuquerque, New Mexico
  - Mount Sinai School Of Medicine, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Dumc, Durham, North Carolina
  - University Hospitals Of Cleveland, Cleveland, Ohio
  - University Hospitals, Cleveland, Ohio

REFERENCES:
- [Derived] Amin A, Lawson DH, Salama AK, Koon HB, Guthrie T Jr, Thomas SS, O'Day SJ, Shaheen MF, Zhang B, Francis S, Hodi FS. Phase II study of vemurafenib followed by ipilimumab in patients with previously untreated BRAF-mutated metastatic melanoma. J Immunother Cancer. 2016 Aug 16;4:44. doi: 10.1186/s40425-016-0148-7. eCollection 2016. PMID 27532019
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 70 patients were enrolled, and 46 received treatment.
Period: Vem 1 Phase (Vemurafenib, 960 mg)
Arm/Group | Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg
Started | 46
Completed | 46
Not Completed | 0
Period: Ipilimumab Phase (Ipilimumab, 10 mg/kg)
Arm/Group | Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg
Started | 46
Completed | 19
Not Completed | 27
Not completed — Disease progression | 7
Not completed — Study drug toxicity | 6
Not completed — Administrative Reason by Sponsor | 2
Not completed — Adverse event unrelated to study drug | 1
Not completed — Maximum clinical benefit | 1
Not completed — Death | 1
Not completed — Not identified | 2
Not completed — Not reported | 7
Period: Vem 2 Phase (Vemurafenib Retreatment)
Arm/Group | Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg
Started | 19
Completed | 0
Not Completed | 19
Not completed — Disease progression | 12
Not completed — Study drug toxicity | 5
Not completed — Adverse event unrelated to study drug | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (14.20)
Age, Continuous [Median (Full Range); unit: Years] | 57.5 [18 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 37
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 42
  Other | 4
M-Stage at Study Entry [Number; unit: Participants] — M-stage=stage of metastases (M), based on criteria of the American Joint Committee on Cancer. M0=no metastases. M1A=metastases to skin, subcutaneous tissue, or distant lymph nodes. M1B=metastases to lung. M1C=metastases to all other visceral sites or distant metastases to any site combined with an elevated serum level of lactase dehydrogenase.
  Participants
    M0 | 6
    M1A | 8
    M1B | 8
    M1C | 24
Disease Stage at Study Entry [Number; unit: Participants] — Melanoma staging criteria: Stage III (A,B,C)=The tumor may be of any thickness and may or may not be ulcerated. The cancer cells have spread either to a few nearby lymph nodes or tissue just outside the tumor but not to the lymph nodes. Stage IV=The cancer cells have spread to the lymph nodes, other organs in the body, or areas far from the original site of the tumor. This is called metastatic melanoma.
  Participants
    III | 8
    IV | 38
Number of Disease Sites [Number; unit: Participants]
  1 | 2
  2 | 8
  3 | 7
  4 | 4
  5 or more | 25
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — ECOG is a 6-item scale used to assess disease progression, daily functioning, and appropriate treatment and prognosis. Performance status is scored on a scale ranging from 0-5, with (best score) 0=fully active and able to carry on all predisease performance without restriction and (worst score) 5=death.
  Participants
    0 | 35
    1 | 11
Time from Diagnosis of Advanced /Metastatic Melanoma to First Vem1 Phase Dose [Mean (Standard Deviation); unit: Months] — Vem=vemurafenib.
  Months | 4.96 (9.38)
Time from Diagnosis of Advanced /Metastatic Melanoma to First Vem1 Phase Dose [Median (Full Range); unit: Months] — Vem=vemurafenib
  Months | 1.86 [0.3 to 52.3]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Received Ipilimumab and Who Had Grade 3-4 Drug-related Skin Adverse Events (AEs)
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Drug-related=having certain, probable, possible, or unknown relationship to study drug. Grading criteria for AEs: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death.
Time Frame: From the first dose date of Vem1 to the last dose of ipilimumab (to a maximum of 3 years) + 90 days or to the first dose date of Vem2, whichever occurred first
Population: All participants who received at least 1 dose of ipilimumab
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg: Participants received vemurafenib, 960 mg, twice daily for 6 weeks (Vem1 Phase). After a washout period of 3-10 days, patients received ipilimumab, 10 mg/kg, every 3 weeks for a maximum of 4 doses. At Week 24, participants received ipilimumab, 10 mg/kg, every 12 weeks until disease progression or unacceptable toxicity. Patients who did not progress or have unacceptable toxicity in the Vem1 Phase were retreated with vemurafenib (Vem 2 Phase) at the last dose level identified at the end of the Vem1 Phase until disease progression or unacceptable toxicity. Following the end-of-treatment visit, patients entered the Follow-up Phase.
Arm/Group | Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg
Number analyzed (Participants) | 46
Percentage of participants | 32.6 [19.5 to 48.0]

2. Secondary Outcome: Percentage of Participants Who Received Ipilimumab and Who Had Grade 3-4 Drug-related Gastrointestinal Adverse Events (AEs)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of ipilimumab.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg
Number analyzed (Participants) | 46
Percentage of participants | 21.7 [10.9 to 36.4]

3. Secondary Outcome: Percentage of Participants Who Received Ipilimumab and Who Had Grade 3-4 Drug-related Hepatobiliary Adverse Events
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of vemurafenib and ipilimumab
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg
Number analyzed (Participants) | 46
Percentage of participants | 4.3 [0.5 to 14.8]

4. Other Pre Specified Outcome: Number of Participants Who Died, Who Died Due to Related Adverse Events (AEs), and With Related AEs, Serious Adverse Events (SAEs), Related SAEs, Discontinuations Due to AEs and Related AEs, Immune-related (ir) AEs, and Serious irAEs
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or unknown relationship to study drug.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg
Number analyzed (Participants) | 46
Participants
  Deaths | 4
  Deaths due to related AEs | 0
  SAEs | 31
  Related SAEs | 18
  Discontinuations due to AEs | 18
  Discontinuations due to related AEs | 16
  irAEs | 43
  Serious irAEs | 10

5. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) Grade 3-4, Related AEs Grade 3-4, Related Serious Adverse Events (SAEs) Grade 3-4, Immune-related (ir) AEs Grade 3-4, and Serious irAEs Grade 3-4
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or unknown relationship to study drug. Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Vemurafenib, 960 mg + Ipilimumab, 10 mg/kg
Number analyzed (Participants) | 46
Participants
  AEs Grade 3-4 | 39
  Related AEs Grade 3-4 | 30
  Related SAEs Grade 3-4 | 17
  irAEs Grade 3-4 | 25
  Serious irAEs Grade 3-4 | 9

ADVERSE EVENTS:
Time Frame: AEs with onset date on or after Day 1 of study therapy and within the last dose of Vem1 + 14 days, last dose of Ipi Phase + 90 days, last dose of Vem2 + 14 days. Up to July 2014 (approximately 21 months)
Groups:
- Vemurafenib, 960 mg + Ipilimumab,10 mg/kg ab: Participants received vemurafenib, 960 mg, twice daily for 6 weeks (Vem1 Phase). After a washout period of 3-10 days, patients received ipilimumab, 10 mg/kg, every 3 weeks for a maximum of 4 doses. At Week 24, participants received ipilimumab, 10 mg/kg, every 12 weeks until disease progression or unacceptable toxicity. Patients who did not progress or have unacceptable toxicity in the Vem1 Phase were retreated with vemurafenib (Vem 2 Phase) at the last dose level identified at the end of the Vem1 Phase until disease progression or unacceptable toxicity.
Arm/Group | Vemurafenib, 960 mg + Ipilimumab,10 mg/kg ab
Serious Adverse Events (participants affected / at risk) | 34/46
Other Adverse Events (participants affected / at risk) | 44/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib, 960 mg + Ipilimumab,10 mg/kg ab (N=46)
Colitis (Gastrointestinal disorders) | 3
Hepatitis (Hepatobiliary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abasia (General disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Iliac vein occlusion (Vascular disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Pancreatitis (Gastrointestinal disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Headache (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Hypotension (Vascular disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pneumonia (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Blood creatine increased (Investigations) | 1
Dysphagia (Gastrointestinal disorders) | 2
Hepatic enzyme increased (Investigations) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Wound (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 1
Hypopituitarism (Endocrine disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyrexia (General disorders) | 2
Adrenal Insufficiency (Endocrine disorders) | 1
Hypophysitis (Endocrine disorders) | 1
Cellulitis (Infections and infestations) | 1
Haemorrhage Intracranial (Nervous system disorders) | 2
Autoimmune Colitis (Gastrointestinal disorders) | 1
Peripheral Swelling (General disorders) | 1
Blood Creatinine Increased (Investigations) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib, 960 mg + Ipilimumab,10 mg/kg ab (N=46)
Blood alkaline phosphatase increased (Investigations) | 11
Colitis (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 9
Dysgeusia (Nervous system disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 4
Flushing (Vascular disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Hyperaesthesia (Nervous system disorders) | 3
Pollakiuria (Renal and urinary disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 31
Vision blurred (Eye disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Blood sodium decreased (Investigations) | 4
Constipation (Gastrointestinal disorders) | 9
Decreased appetite (Metabolism and nutrition disorders) | 19
Headache (Nervous system disorders) | 15
Hypokalaemia (Metabolism and nutrition disorders) | 8
Mucosal inflammation (General disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7
Adrenal insufficiency (Endocrine disorders) | 3
Blood calcium decreased (Investigations) | 4
Blood creatinine increased (Investigations) | 8
Dizziness (Nervous system disorders) | 11
Erythema (Skin and subcutaneous tissue disorders) | 4
Exfoliative rash (Skin and subcutaneous tissue disorders) | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Lipase increased (Investigations) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Urinary tract infection (Infections and infestations) | 5
Vomiting (Gastrointestinal disorders) | 16
Candida infection (Infections and infestations) | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 23
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hypothyroidism (Endocrine disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Pain (General disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 19
Weight decreased (Investigations) | 5
Anxiety (Psychiatric disorders) | 3
Hot flush (Vascular disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 6
Hypophysitis (Endocrine disorders) | 7
Oedema peripheral (General disorders) | 11
Sinusitis (Infections and infestations) | 4
Abdominal pain (Gastrointestinal disorders) | 13
Alopecia (Skin and subcutaneous tissue disorders) | 7
Aspartate aminotransferase increased (Investigations) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 11
Chills (General disorders) | 10
Dysphagia (Gastrointestinal disorders) | 5
Hypertension (Vascular disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Insomnia (Psychiatric disorders) | 14
Nausea (Gastrointestinal disorders) | 22
Night sweats (Skin and subcutaneous tissue disorders) | 3
Alanine aminotransferase increased (Investigations) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Fatigue (General disorders) | 24
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 7
Lymphocyte count decreased (Investigations) | 3
Pyrexia (General disorders) | 14
Cellulitis (Infections and infestations) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.